CLINICAL TRIAL: NCT02160821
Title: Transversus Abdominis Plane Block Versus Caudal Epidural for Lower Abdominal Surgery in Children: A Double-Blinded Randomized Controlled Trial
Brief Title: TAPB vs. Caudal for Lower Abdominal Surgery in Children: A Double-Blinded Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1610841001
Record Dates: First submitted 2014-05-29; First posted 2014-06-11 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Anesthesia, Recovery Period
Keywords: Transversus Abdominis Plane Block; Caudal Epidural; Pediatric Pain control; Pain control for Lower Abdominal Surgery
MeSH Terms: interventions — Anesthesia, Caudal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transversus Abdominis Plane Block (Experimental): Transversus Abdominis Plane Block TAPB Ultrasound guided TAPB
  Interventions: Procedure: Transversus Abdominis Plane Block
- Caudal Epidural Block (Experimental): Caudal Epidural Block Caudal Block Neuraxial Block Ultrasound Guided Caudal Block
  Interventions: Procedure: Caudal Epidural

INTERVENTIONS:
Procedure: Caudal Epidural — Ultrasound Guided Caudal Block
  Arms: Caudal Epidural Block
Procedure: Transversus Abdominis Plane Block — Ultrasound Guided Transversus Abdominis Plane Block
  Arms: Transversus Abdominis Plane Block

SUMMARY:
Transversus abdominis plane block (TAPB) has emerged as a safe and effective regional anesthesia technique for providing postoperative lower abdominal analgesia. Complications associated with TAPB are very rare and pose a lower overall risk to the patient receiving a TAPB versus a caudal block, which is considered the gold standard for pediatric lower abdominal regional anesthesia. Our study hypothesis was that TAPB would be equivalent to caudal block initially in providing postoperative pain control but would show improved pain relief beyond the anticipated caudal duration.

DETAILED DESCRIPTION:
The study design was a double-blinded randomized controlled trial. A minimum of 44 children between the ages of 1 and 9 undergoing bilateral ureteral reimplantation surgery through a low transverse incision will be enrolled. Narcotic requirement, pain scores (FLACC/FACES), episodes of nausea/vomiting, and anti-spasmodic requirement will be recorded in the PACU and at 6 hour intervals through 24 hours from the time of the block placement.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 1 to 9 years old scheduled for intravesicular ureteral reimplantation surgery

Exclusion Criteria:

1. Coagulation status or anatomic variations precluded safe placement of either TAPB or caudal epidural,
2. there was a preexisting chronic pain disorder,
3. there was a history of constipation that persisted despite appropriate treatment and that may have impacted postoperative pain assessments,
4. additional procedures were planned via a separate incision at the time of the ureteral reimplantation, 5) there was a contraindication to receiving the medications described in the protocol.

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2011-01; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Narcotic requirement | 24 hours post intervention
  Narcotic requirement was recorded at 24 hours from the time of the block placement.

SECONDARY OUTCOMES:
episodes of nausea/vomiting | 24 hours
  Episodes of nausea/vomiting were recorded at 24 hours from the time of the block placement.
anti-spasmodic requirement | 24 hours post intervention
  Anti-spasmodic requirement were recorded at 24 hours from the time of the block placement.
Pain Scores | 24 hours post intervention
  Pain scores (FLACC/FACES) were recorded at 24 hours from the time of the block placement

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Bryskin, MD, Principal Investigator — Nemours Children's Clinic
Locations (1):
- Wolfson Children's Hospital, Baptist Medical Center- Downtown, 800 Prudential Drive, Jacksonville, Florida, United States

REFERENCES:
- [Background] Tripi PA, Palmer JS, Thomas S, Elder JS. Clonidine increases duration of bupivacaine caudal analgesia for ureteroneocystostomy: a double-blind prospective trial. J Urol. 2005 Sep;174(3):1081-3. doi: 10.1097/01.ju.0000169138.90628.b9. PMID 16094063
- [Background] Vetter TR, Carvallo D, Johnson JL, Mazurek MS, Presson RG Jr. A comparison of single-dose caudal clonidine, morphine, or hydromorphone combined with ropivacaine in pediatric patients undergoing ureteral reimplantation. Anesth Analg. 2007 Jun;104(6):1356-63, table of contents. doi: 10.1213/01.ane.0000261521.52562.de. PMID 17513626
- [Derived] Bryskin RB, Londergan B, Wheatley R, Heng R, Lewis M, Barraza M, Mercer E, Ye G. Transversus Abdominis Plane Block Versus Caudal Epidural for Lower Abdominal Surgery in Children: A Double-Blinded Randomized Controlled Trial. Anesth Analg. 2015 Aug;121(2):471-8. doi: 10.1213/ANE.0000000000000779. PMID 25902326